CLINICAL TRIAL: NCT04297202
Title: A Phase II, Open-label, Single Arm, Investigator-initiated Trail of An Anti-PD-1 Inhibitor SHR-1210 in Combination With Apatinib in the Perioperative Treatment of Hepatocellular Carcinoma
Brief Title: SHR-1210 Combined With Apatinib Mesylate in the Perioperative Treatment of Hepatocellular Carcinoma
Acronym: HCC-009
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: The First Affiliated Hospital with Nanjing Medical University (Other)
Collaborators: Jiangsu Hengrui Pharmaceutical Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2019-SR-332
Record Dates: First submitted 2020-01-30; First posted 2020-03-05 (Actual); Last update posted 2020-08-07 (Actual); Status verified 2020-08

CONDITIONS: Hepatocellular Carcinoma
Keywords: Hepatocellular Carcinoma; the Perioperative Treatment; HCC
MeSH Terms: conditions — Carcinoma, Hepatocellular | interventions — camrelizumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Apatinib Combined With SHR-1210 Injection (Experimental): SHR-1210 Injection: 3 cycles of neoadjuvant therapy before surgery, two weeks is a treatment cycle; Apatinib : D1-D21 : 250 mg, orally, qd; Before surgery, the patient's surgical pathology samples still need to be collected.
  D46 : Patients were preoperatively evaluated. Operable patients were scheduled for hepatectomy with/without microwave ablation;
  After 4 to 8 weeks after liver resection, a postoperative adjuvant program is performed. The cycle of a three-week plan will be performed with a total of 8 cycles with the treatment of Apatinib combination with SHR-1210 Injection.
  Interventions: Drug: Apatinib Combined With SHR-1210 Injection

INTERVENTIONS:
Drug: Apatinib Combined With SHR-1210 Injection — 3 cycles of neoadjuvant therapy before surgery, two weeks is a treatment cycle: D1、D15、D31 : SHR-1210 200mg, I.V, q2w； D1-D20 : Apatinib 250 mg, orally, qd; D46 : Patients were preoperatively evaluated. Operable patients were scheduled for hepatectomy with/without microwave ablation; After 4 to 8 weeks after liver resection, a postoperative adjuvant program is performed. Three weeks is a treatment cycle with a total of 8 cycles
  In each cycle:
  D1: SHR-1210 200mg, I.V, q3w; D1-D21: Apatinib 250mg, orally, qd;

SUMMARY:
This is a Phase II , Open-label , Investigator-initiated Trail of SHR-1210 (an Anti-PD-1 Inhibitor) in Combination With Apatinib in Patients With Hepatocellular Carcinoma(HCC).This study aims to evaluate the safety and efficacy of SHR-1210 combination with Apatinib as a preoperative treatment of HCC.

DETAILED DESCRIPTION:
This is an Open, Single Arm, Exploratory and Phase II Clinical Trial of Apatinib Combined With SHR-1210 (an Anti-PD-1 Inhibitor) in Patients With Hepatocellular Carcinoma(HCC) as Perioperative Treatment. we conduct this study in order to observe and evaluate the efficacy and safety of Apatinib combined with SHR-1210 (an Anti-PD-1 Inhibitor) in treatment of patients with HCC. Primary Efficacy Endpoint: Major pathologic response (MPR), Secondary Efficacy Endpoints: Pathological complete response Rate (pCR), Objective Response(ORR) (According to RECIST Version 1.1), Recurrence-free survival(RFS) and Overall survival rate of 6 months (OS %-6 m). Safety and tolerance will be evaluated by incidence, severity and outcomes of AEs and categorized by severity in accordance with the NCI CTC AE Version 4.0.3.

ELIGIBILITY:
Inclusion Criteria:

1. The patient volunteered to participate in the study and signed an informed consent form
2. ≥18 years of age，Male or female
3. Subjects are diagnosed with histologically or cytologically confirmed HCC
4. Subjects haven't received any systemic treatment for HCC before admission.
5. Subjects enrolled must have measurable lesion(s) according to the RECIST 1.1 standard
6. ECOG performance status of 0 or 1
7. Life expectancy ≥ 12 weeks
8. Subjects are diagnosed with resectable stage IIB, stage IIIA HCC cancer.
9. The main organ's function is normal and it should meet the following criteria(Excludes use of any blood components and cell growth factors during the screening period)

   1. Absolute neutrophil count≥1.5×109 /L
   2. Platelets≥80×109/L ;Hemoglobin≥9.0 g/dL; Serum albumin≥3g/dL
   3. Thyroid stimulating hormone (TSH)≤1.0×upper limit of normal(ULN)（If abnormal, T3 and T4 levels should be examined at the same time）
   4. Total bilirubin (TBIL)≤1.5×upper limit of normal (ULN); ALT and AST≤1.5×upper limit of normal(ULN); AKP≤ 2.5×upper limit of normal(ULN)
   5. Serum creatinine ≤1.5×ULN or creatinine clearance > 60 mL/minute (using Cockcroft-Gault formula)

Exclusion Criteria:

1. Known hepatocholangiocarcinoma, sarcomatoid HCC, mixed cell carcinoma and lamellar cell carcinoma; other active malignant tumor except HCC within 5 years or simultaneously
2. Be ready for or previously received organ or allogenic bone marrow transplantation
3. Moderate-to-severe ascites with clinical symptoms
4. History of gastrointestinal hemorrhage within 6 months prior to the start of study treatment or clear tendency of gastrointestinal hemorrhage.
5. Abdominal fistula, gastrointestinal perforation or intraperitoneal abscess within 6 months prior to the start of study treatment.
6. Known genetic or acquired hemorrhage or thrombotic tendency.
7. The patient is currently using or has recently used (within 10 days before the start of study treatment) aspirin (> 325mg / day (maximum antiplatelet dose) or dipyridamole, ticlopidine, clopidogrel and cilostazol.
8. Thrombosis or thromboembolic event within 6 months prior to the start of study treatment.
9. Cardiac clinical symptom or disease that is not well controlled.
10. Subjects have uncontrollable hypertension (systolic pressure ≥ 140 mmHg or diastolic pressure ≥ 90 mmHg), despite patients have taken the best drug treatment ；Subjects have had a hypertensive crisis or hypertensive encephalopathy
11. Patient develops severe vascular disease within 6 months before the start of study treatment.
12. Patients with severe, unhealed or split wounds and active ulcers or untreated fractures
13. Patients who underwent surgical treatment within 4 weeks prior to the start of study treatment.
14. Factors to affect oral administration (such as patients unable to swallow oral medications, malabsorption syndrome etc. situations evidently affect drug absorption).
15. Patients with gastrointestinal diseases such as intestinal obstruction (including incomplete intestinal obstruction) or those who may have caused gastrointestinal bleeding, perforation or obstruction.
16. There is evidence of intragastric gas that cannot be explained by puncture or recent surgery.
17. Previous or current presence of metastasis to central nervous system.
18. Subjects have history of hepatic encephalopathy.
19. The subject has an interstitial lung disease that is symptomatic or may interfere with the discovery or management of suspected drug-related lung toxicity; previous and current subjects with a history of pulmonary fibrosis, interstitial pneumonia, pneumoconiosis, drug-associated pneumonia, severe impaired lung function, etc.
20. The patient has any active autoimmune disease or a history of autoimmune disease expected relapse.
21. Severe infection within 4 weeks prior to the start of study treatment.
22. A history of immunodeficiency, including HIV-positive or other acquired, congenital immunodeficiency disease.
23. Prior therapy with any anti-PD-1/PD-L1 drug (specifically targeting T-cell co-stimulation or checkpoint pathways), Sorafenib or Apatinib.
24. Subjects were vaccinated with live attenuated vaccine within 28 days before the first dose or expected to receive this vaccine within 60 days after the last dose or during the study period.
25. Treatment of other investigational product(s) within 28 days prior to the start of study treatment.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 20 (Estimated)
Dates: Start 2019-12-01 (Actual); Primary Completion 2021-12-01 (Estimated); Study Completion 2021-12-01 (Estimated)

PRIMARY OUTCOMES:
Major pathologic response | 6 months
  It is defined as residual tumors less than 10% after neo-adjuvant therapy

SECONDARY OUTCOMES:
Pathological complete response | 6 months
  No histologic evidence of malignancy or only the ingredients of carcinoma in situ was found in primary tumors
Objective Response(ORR) | Before surgery；
  It is defined as the proportion of patients whose tumors shrink to a predetermined size and maintain a minimum time limit. It includes the cases of CR and PR.
Recurrence free survival(RFS) | through study completion, an average of 1 year
  from surgery to relapse or death resulting from any cause .
Recurrence free survival rates of 6 months and 12 months | 12 months
  the rate of proportion of all patients from surgery to relapse or death resulting from any cause.
Overall survival rate (6 m or 12 m) | through study completion; the rate of OS for 6 months and 12 months
  It is defined as the time from randomization to death from any cause during the course of the study
Safety as measured by the rate of AEs | through study completion, an average of 1 year
  Safety will be evaluated by incidence, severity and outcomes of adverse events (AEs) and categorized by severity in accordance with the NCI CTC AE Version 4.0.3

CONTACTS AND LOCATIONS:
Overall Officials: Xuehao Wang, Study Chair — The First Affiliated Hospital with Nanjing Medical University
Locations (1):
- Jiangsu Province Hospital, Nanjing, Jiangsu, China

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Xia Y, Tang W, Qian X, Li X, Cheng F, Wang K, Zhang F, Zhang C, Li D, Song J, Zhang H, Zhao J, Yao A, Wu X, Wu C, Ji G, Liu X, Zhu F, Qin L, Xiao X, Deng Z, Kong X, Li S, Yu Y, Xi W, Deng W, Qi C, Liu H, Pu L, Wang P, Wang X. Efficacy and safety of camrelizumab plus apatinib during the perioperative period in resectable hepatocellular carcinoma: a single-arm, open label, phase II clinical trial. J Immunother Cancer. 2022 Apr;10(4):e004656. doi: 10.1136/jitc-2022-004656. PMID 35379737